CLINICAL TRIAL: NCT02975206
Title: A Randomized, Double-Blind, Placebo Controlled Study Of The Efficacy, Safety, And Tolerability Of Serlopitant For The Treatment Of Pruritus In Adults And Adolescents With A History Of Atopic Dermatitis
Brief Title: Study of the Efficacy, Safety, and Tolerability of Serlopitant for Pruritus (Itch) in Atopic Dermatitis
Acronym: ATOMIK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTI-103
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Pruritus; Atopic Dermatitis
MeSH Terms: conditions — Pruritus; Dermatitis, Atopic | interventions — serlopitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Serlopitant High Dose (Experimental): serlopitant tablets - high dose
  Interventions: Drug: Serlopitant High Dose
- Serlopitant Low Dose (Experimental): serlopitant tablets - low dose
  Interventions: Drug: Serlopitant Low Dose
- Placebo Oral Tablet (Placebo Comparator): matching placebo tablets
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Serlopitant High Dose — serlopitant tablets - high dose
  Arms: Serlopitant High Dose
Drug: Placebo Oral Tablet — placebo tablet
  Arms: Placebo Oral Tablet
Drug: Serlopitant Low Dose — serlopitant tablets - low dose
  Arms: Serlopitant Low Dose

SUMMARY:
Study of the Efficacy, Safety, and Tolerability of Serlopitant for Pruritus (Itch) in Atopic Dermatitis

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled study. Approximately 450 subjects will be randomized in a 1:1:1 ratio to receive daily oral doses of serlopitant 1 mg, 5 mg, or placebo for 6 weeks. During the screening period, subjects will be provided with an electronic device for recording electronic diary (eDiary) assessments throughout the study. This eDiary will be used to capture efficacy endpoint data and treatment information. At the Baseline visit, eligible subjects will be randomized, and study drug dispensed beginning with a loading dose of 3 tablets to be taken at bedtime that same day. Starting on Study Day 2, subjects will take one tablet per day at bedtime. Treatment will continue for 6 weeks. The primary efficacy endpoint will be assessed during Week 6. After completion of the 6-week treatment period, all subjects will enter a 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 13 years or older
* Pruritus prior to and during the initial screening period
* Diagnosis of atopic dermatitis
* Judged to be in good health in the investigator's opinion

Exclusion Criteria:

* Prior treatment with study drug or similar drug
* Pruritus due to another reason besides atopic dermatitis
* Presence of any medical condition or disability that could interfere with study
* History of hypersensitivity to serlopitant or any of its components
* Currently pregnant or male partner of pregnant female
* Females of childbearing potential who are unable or unwilling to use adequate contraception or who are breast feeding

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Spellman, MD, Study Director — Vyne Therapeutics Inc.
Locations (52):
- United States (52):
  - Study Site 332, Anniston, Alabama
  - Study Site 363, Birmingham, Alabama
  - Study Site 340, Hoover, Alabama
  - Study Site 364, Glendale, Arizona
  - Study Site 334, Cerritos, California
  - Study Site 386, Encinitas, California
  - Study Site 366, Fountain Valley, California
  - Study Site 338, Los Angeles, California
  - Study Site 383, North Hollywood, California
  - Study Site 374, Oceanside, California
  - Study Site 347, San Diego, California
  - Study Site 356, San Diego, California
  - Study Site 333, San Francisco, California
  - Study Site 376, Santa Monica, California
  - Study Site 358, Denver, Colorado
  - Study Site 370, Jacksonville, Florida
  - Study Site 331, Miami, Florida
  - Study Site 348, Miami, Florida
  - Study Site 378, Miami, Florida
  - Study Site 353, Pinellas Park, Florida
  - Study Site 368, Tampa, Florida
  - Study Site 377, Tampa, Florida
  - Study Site 369, Atlanta, Georgia
  - Study Site 349, Savannah, Georgia
  - Study Site 381, Chicago, Illinois
  - Study Site 360, New Albany, Indiana
  - Study Site 380, Bardstown, Kentucky
  - Study Site 344, Louisville, Kentucky
  - Study Site 379, Boston, Massachusetts
  - Study Site 350, Warren, Michigan
  - Study Site 371, Saint Joseph, Missouri
  - Study Site 387, Las Vegas, Nevada
  - Study Site 352, Berlin, New Jersey
  - Study Site 375, Forest Hills, New York
  - Study Site 373, Rochester, New York
  - Study Site 341, High Point, North Carolina
  - Study Site 355, Shelby, North Carolina
  - Study Site 337, Oklahoma City, Oklahoma
  - Study Site 345, Johnston, Rhode Island
  - Study Site 362, Providence, Rhode Island
  - Study Site 382, Anderson, South Carolina
  - Study Site 343, Spartanburg, South Carolina
  - Study Site 357, Chattanooga, Tennessee
  - Study Site 365, Austin, Texas
  - Study Site 335, Houston, Texas
  - Study Site 359, Pflugerville, Texas
  - Study Site 339, Plano, Texas
  - Study Site 361, San Antonio, Texas
  - Study Site 351, Draper, Utah
  - Study Site 342, Norfolk, Virginia
  - Study Site 336, Richmond, Virginia
  - Study Site 367, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Serlopitant 5 mg: Subjects received a 3-tablet oral loading dose on the first day of the treatment period followed by an oral 5 mg dose of Serlopitant taken once daily by mouth for 6 weeks
- Serlopitant 1 mg: Subjects received a 3-tablet oral loading dose on the first day of the treatment period followed by an oral 1 mg dose of Serlopitant taken once daily by mouth for 6 weeks
- Placebo Oral Tablet: Subjects received a 3-tablet oral loading dose on the first day of the treatment period followed by an oral Placebo tablet taken once daily by mouth for 6 weeks
Period: Overall Study
Arm/Group | Serlopitant 5 mg | Serlopitant 1 mg | Placebo Oral Tablet
Started | 161 | 161 | 162
Completed | 134 | 144 | 145
Not Completed | 27 | 17 | 17
Not completed — Withdrawal by Subject | 14 | 11 | 11
Not completed — Other (e.g., lost to follow up) | 13 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Placebo Oral Tablet: Subjects received a 3-tablet Placebo oral loading dose on the first day of the treatment period followed by an oral Placebo tablet taken once daily by mouth for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Serlopitant 5 mg | Serlopitant 1 mg | Placebo Oral Tablet | Total
Number analyzed (Participants) | 161 | 161 | 162 | 484
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 15 | 10 | 45
  Between 18 and 65 years | 131 | 138 | 149 | 418
  >=65 years | 10 | 8 | 3 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (16.62) | 38.1 (15.16) | 37.5 (13.04) | 37.1 (15.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 109 | 108 | 325
  Male | 53 | 52 | 54 | 159
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 22 | 18 | 19 | 59
  Race: Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 4
  Race: Black or African American | 64 | 67 | 69 | 200
  Race: White | 69 | 70 | 68 | 207
  Race: More than one race | 2 | 3 | 2 | 7
  Race: Unknown or Not Reported | 2 | 2 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 161 | 161 | 162 | 484
WI-NRS [Mean (Standard Deviation); unit: units on a scale] — Worst Itch Numeric Rating Scale (WI-NRS). 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. Subject-reported score from reflection on past 24 hours. The baseline was established by averaging 7 daily scores leading up to randomization. Population: The row populations here represent the Full Analysis Set, not all subjects randomized.
  units on a scale
    number analyzed (Participants) | 160 | 161 | 158 | 479
    (all) | 8.38 (0.993) | 8.23 (1.039) | 8.26 (1.057) | 8.29 (1.029)

OUTCOME MEASURES:

1. Primary Outcome: Change in WI-NRS From Baseline to Week 6
Description: Worst Itch Numeric Rating Scale (WI-NRS). 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. The primary outcome is the change in WI-NRS score between the visit and Baseline.
Time Frame: Week 6 compared to Baseline
Population: These figures represent full analysis set.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo Oral Tablet: Subjects received a 3-tablet oral loading dose on the first day of the treatment period followed by an oral Placebo taken once daily by mouth for 6 weeks
Arm/Group | Serlopitant 5 mg | Serlopitant 1 mg | Placebo Oral Tablet
Number analyzed (Participants) | 160 | 161 | 158
score on a scale | -2.25 (2.198) | -2.32 (2.418) | -2.01 (2.212)

2. Secondary Outcome: WI-NRS 4-point Responder Rate at Week 6
Description: Worst Itch Numeric Rating Scale (WI-NRS). 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. A 4-point responder is a subject who had at least a 4-point reduction in score between Week 6 and baseline.
Time Frame: Week 6 compared to Baseline
Population: These figures represent full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Serlopitant 5 mg | Serlopitant 1 mg | Placebo Oral Tablet
Number analyzed (Participants) | 160 | 161 | 158
Participants | 33 | 36 | 26

3. Secondary Outcome: Change in Quality of Life (ItchyQoL) From Baseline to Week 6
Description: ItchyQoL is a 22-item pruritus-specific instrument that measures the degree to which pruritus affects quality-of-life. The responses to the items are Never (1), Rarely (2), Sometimes (3), Often (4) and All the Time (5). A higher score corresponds to a more adverse impact. The overall score is the average of the 22 items ranging from 1 to 5.
Time Frame: Week 6 compared to Baseline
Population: These figures represent all participants in the full analysis set who completed the ItchyQol assessment at both Baseline and Week 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Serlopitant 5 mg | Serlopitant 1 mg | Placebo Oral Tablet
Number analyzed (Participants) | 130 | 142 | 139
score on a scale | -0.57 (0.749) | -0.58 (0.779) | -0.53 (0.683)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were recorded from the first study drug administration through the follow-up visit at Week 10. After the Week 10 visit, SAEs that are believed to be drug related will be reported, without a specific end time.
Description: The at risk safety population is a subset of participants who received at least one dose of study medication. This population is analyzed based upon the actual treatment received, at the highest dose received.
Arm/Group | Serlopitant 5 mg | Serlopitant 1 mg | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 1/161 | 0/160 | 0/158
Serious Adverse Events (participants affected / at risk) | 2/161 | 1/160 | 2/158
Other Adverse Events (participants affected / at risk) | 27/161 | 22/160 | 32/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serlopitant 5 mg (N=161) | Serlopitant 1 mg (N=160) | Placebo Oral Tablet (N=158)
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Serlopitant 5 mg (N=161) | Serlopitant 1 mg (N=160) | Placebo Oral Tablet (N=158)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 9 | 2 | 5
Urinary tract infection (Infections and infestations) | 5 | 5 | 4
Nasopharyngitis (Infections and infestations) | 6 | 2 | 5
Headache (Nervous system disorders) | 2 | 2 | 5
Somnolence (Nervous system disorders) | 2 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT02975206/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT02975206/SAP_001.pdf